CLINICAL TRIAL: NCT06824038
Title: Impact of Nutrition Counseling on the Nutritional Status of Patients With Ulcerative Colitis: A Randomized Controlled Clinical Trial
Brief Title: Nutritional Counseling Impact on Ulcerative Colitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rahma Mohammed Medhat Ali (Other)
Responsible Party: Sponsor-Investigator, Rahma Mohammed Medhat Ali, assistant lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MD-53-2023
Record Dates: First submitted 2025-01-29; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): Patients with moderate Ulcerative Colitis, in active phase, Ages: Adults aged 18-60, of both sexes. Intervention: will receive nutritional counseling sessions ,nd weekly follow-up through clinic vists and mobile phones and messaging
  Interventions: Behavioral: nutritional counseling
- control group (No Intervention): Patients with moderate Ulcerative Colitis, in active phase. Adults aged 18-60, of both sexes.
  will receive regular care of the clinic.

INTERVENTIONS:
Behavioral: nutritional counseling — Nutritional counseling based on the nutritional assessment of each patient. Each patient will receive a package of:
  i. A booklet that contains the whole instructions and dietary records to help in remembering information and record their application of the plan.
  ii. A tailored diet menu adjusted according to the required calories of the patient calculated by the Harris Benedict equation, considering the patient preferences, individualized requirements and with choices suitable for different economic classes.
  Arms: intervention group

SUMMARY:
randomized clinical trial aimed to find whether, In ulcerative colitis patients, nutrition counseling is associated with improved nutritional status.

objectives:

1. Asses the nutritional status and quality of life among a sample of UC patients attending the NHTMRI outpatient clinic.
2. Provide nutritional counseling for the randomly allocated intervention group
3. Evaluate the effect of the nutritional counseling on nutritional status, quality of life and disease progression.

   * Inclusion criteria: patients with moderate Ulcerative Colitis, in active phase. Adults aged 18-60, of both sexes

Patients in the intervention group will receive a counseling session then instructs on the subsequent follow up dates. Each patient of the intervention group is scheduled to receive weekly session, according to settled appointments; while the control arm will receive the regular service at the clinic.

DETAILED DESCRIPTION:
Administrative and Preparatory Phase:

After obtaining approval from the corresponding parties, a booklet in Arabic language with educational material and instruction will be prepared. Common foods for and against bowel discomfort will be emphasized. Dietary records will be included to check the adherence of the patients to the instructions.

II- Pre-intervention phase (The initial assessment):

The investigator will review the medical record of each patient to confirm the diagnosis and severity; then eligible patients in both counseling arm and the control arm will be interviewed by the investigator using a structured questionnaire to gather the following data for the initial assessment Personal and socio-demographic data: Comprised enquiry about each patient's age, sex, marital status, occupation, education, residency and telephone/mobile number.

b. Assessment of the quality of life using the short inflammatory bowel disease questionnaire (SIBDQ). It is a set of generic, coherent, and easily administered quality of life measures. Scores are from 0 to 10. A higher score indicates better health.

c. Assessment of the nutritional status by: i. Weight measurement using the German Beurer Glass Scale model GS11 (with large LCD display (digit zone: 25 mm), loading capacity 150 kg and graduation 100 g ii. Height measurement using the Indian wall mounted DESCO stature meter (Model HSHA 101) with a movable horizontal headboard. Maximal height of measuring is 2 m and measurement resolution of 0.5 cm .

iii. Screening all included patients using Nutritional risk screening (NRS 2002). It includes pre-screening with four questions:

1. Is the BMI of the patient < 20.5 kg/m2
2. Did the patient lose weight in the past 3 months?
3. Was the patient's food intake reduced in the past week?
4. Is the patient critically ill? If one of these is answered positively, a screening follows which includes surrogate measures of nutritional status, with static and dynamic parameters and data on the severity of the disease (stress metabolism). For each parameter, a score from 0 to 3 can result. Age over 70 years is considered as a risk factor, and is included in the screening tool as well, giving 1 point. A total score of ≥3 points means that the patient is at risk of malnutrition or already malnourished and therefore a nutritional therapy is indicated.

iv. Handgrip strength (HGS) is a simple and reliable measurement of maximum voluntary muscle strength. It is an important tool for diagnosing sarcopenia and is widely used as a single indicator to represent overall muscle strength, HGS can the incidence of chronic diseases, nutritional status, quality of life, independence of daily life, length of hospital stay, and even mortality v. Skin fold thickness: to measure the double fold of skin and subcutaneous fat to the nearest millimeter. A variety of sites have been used for skinfold measurement, but the most common are triceps, biceps, subscapular and suprailiac.

vi. Assessment of nutritional intake using:

1. Dietary habits questionnaire: The dietary habits questionnaire included enquiry about the number of meals per day, the main meal, breakfast intake, outdoor fatty meals intake, types of snacks, method of cooking meat, method of cooking vegetables, types of fats used in cooking, sports or physical training, sedentary habits, exposure to sun, dietary supplement intake, dietary habits changes during relapse of the disease (relapse duration in days, the number of meals per day, method of cooking meat, method of cooking vegetables)
2. Twenty-four hours dietary recall: The 24-hour dietary recall is an open-ended enquiry about foods consumed during the last 24 hours. It is conducted in an in-depth interview that typically requires 20 to 30 minutes to be completed. Detailed data about food preparation, ingredients in mixed dishes, and the brand name of different commercial products will be collected. Estimation of the amounts of each food consumed in reference to a common size container (e.g., bowls, cups, and glasses), standard measuring cups and spoons. The inevitable limitation is that all information depends on the participants' memory. (Shim et al., 2014) vii) Laboratory assessment: Measurement of Complete blood picture (CBC), and iron.

III- Intervention (Only for the intervention group):

Patients in the intervention group will receive a counseling session then instructs on the subsequent follow up dates. Apart from counseling, patients will receive the same care from the clinic medical staff. After the final assessment, the control group will receive the nutritional counseling material to gain its expected benefits.

Each patient of the intervention group is scheduled to receive weekly session, according to settled appointments. The first session for counseling, the second and the third to check the adherence of the patient to the nutrition plan and to answer any question of the patients as follows:

Session 1: Nutritional counseling based on the nutritional assessment of each patient. Each patient will receive a package of:

i. A booklet that contains the whole instructions and dietary records to help in remembering information and record their application of the plan.

ii. A tailored diet menu adjusted according to the required calories of the patient calculated by the Harris Benedict equation (Habek et al., 2010) considering the patient preferences, individualized requirements and with choices suitable for different economic classes.

Patients will be guided to a diet rich in iron, vitamin D, n-3 fatty acids, and zinc.

Protein requirement are increased in active IBD, and intake should be increased (to 1.2-1.5 g/kg/d in adults) relative to that recommended in the general population.

Probiotic as Lactobacilli can be considered for use in patients with mild to moderate UC for the induction of remission. (Bischoff et al., 2020) A WhatsApp group will be created to add patients at the session 1. Messages will be sent to the patients through the group to stimulate patient adherence to the diet and to remind them of their follow up and final assessment appointments.

Session 2: follow up and reemphasize the instruction. Each patient in the intervention group will receive a weekly telephone follow up session (Tele-health) from a clinical nutritionist to check compliance and respond to inquiries. Between phone sessions, patients can contact their physicians by email or telephone, in addition to the WhatsApp group, or through their routine follow up visits to the IBD clinic to receive their treatment.

I- Post-intervention phase (The final assessment):

All patients in the counseling group and the control groups will be interviewed by the investigator 3 months after the initial assessment session to gather the following data using the same tools of the initial assessment (clinical sheet, follow up laboratory investigations, SIBDQ, NRS 2002, BMI, SFT, HGS, 24 hours dietary recall and dietary habits questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate Ulcerative Colitis, in active phase.
* Adults aged 18-60, of both sexes

Exclusion Criteria:

* Patients with acute fulminant colitis.
* Patient with weight loss > 5% in the last month, and >10% weight loss in the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
nutritional status | three months
  weight in kilograms ,
nutritional status | three months
  body mass index in kg/meter square.
nutritional status | three months
  Nutritional risk screening: The NRS-2002 score is a sum of the total of the nutritional score, severity of disease score and the age adjustment score. The total number of points ranges from 0 to 7. Patients with a score of 3 and more are suggested to have problems with nutrition.
nutritional status | three months
  Hand grip strength measured in kilograms.
nutritional status | three months
  Skin fold thickness in millimeters.
dietary habits | three months
  Dietary habits questionnaire to asses the cooking methods and daily habits.
dietary habits | three months
  Dietary habits questionnaire to asses the cooking methods and daily habits, and, The 24 hour recall to asses food groups intake, macro and micronutrients consumption.
dietary habits | three months
  The 24 hour recall to asses food groups intake, macro and micronutrients consumption.
quality of life score | three months
  asses the QoL through the Short Inflammatory Bowel Disease Questionnaire SIBDQ score. It consists of 10 questions. Each question is scored by a 7-point Likert scale, ranging from 1 (a severe problem) to 7 (not a problem at all), giving an absolute SIBDQ score ranging from 10 (poor health related quality of life "HRQoL") to 70 (optimal HRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Rahma M Ali, Msc, Principal Investigator — Faculty of medicine, Port Said University; Maha A Al Ghobashy, MD, Study Director — Cairo University; Marwa R Salem, MD, Study Director — Cairo University; Kamal A El Atrebi, MD, Study Chair — National hepatology and tropical medicine research institute; Mona Hegazy, MD, Study Chair — Cairo University
Locations (1):
- National Hepatology and Tropical Medicine research institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dryden GW, Dryden SM. Synergistic Benefits of Dietary Strategies in the Management of IBD. Curr Gastroenterol Rep. 2025 Dec;27(1):8. doi: 10.1007/s11894-024-00949-1. Epub 2024 Dec 19. PMID 39702516
- [Background] Jaramillo AP, Abaza A, Sid Idris F, Anis H, Vahora I, Moparthi KP, Al Rushaidi MT, Muddam M, Obajeun OA. Diet as an Optional Treatment in Adults With Inflammatory Bowel Disease: A Systematic Review of the Literature. Cureus. 2023 Jul 18;15(7):e42057. doi: 10.7759/cureus.42057. eCollection 2023 Jul. PMID 37601990